CLINICAL TRIAL: NCT04193020
Title: Impact of Lifestyle and Treatment on the Recurrency and Severity of Acute and Chronic Inflamatory Eye Diseases: Protocol on Prospective Cohort Study
Brief Title: Acute and Chronic Inflammatory Disease, Lifestyle and Treatment Response
Acronym: ACID LTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Principal Investigator, Joanna Przeździecka-Dołyk, Principal Investigator, Wroclaw Medical University
Other Study IDs: ST-859
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- steroid only group (SG)
  Interventions: Other: Surveillance card
- combined (steroid and adjuvant drug) group (CG)
  Interventions: Other: Surveillance card
- bilogic therapy group (BTG)
  Interventions: Other: Surveillance card

INTERVENTIONS:
Other: Surveillance card — Surveillance card and additional examination to find novel markers and better assess the existing ones

SUMMARY:
Acute and chronic inflammatory eye diseases are difficult to diagnose and maintain quiescent with therapy. Proposed study is aimed to find on the one hand, novel factors for recurrence of the disease or remission of inflammation and evaluation of the impact of lifestyle and known factors on the other.

Each patient is treated in accordance to the best of medical knowledge and guidelines for each disease.

This prospective cohort study will enroll uveitic patients to the steroid only group (SG), combined (steroid and adjuvant drug) group (CG) or bilogic therapy group (BTG).

At baseline, patient data are recorded using patient-reported outcome measures and clinical assessments (ophthalomology) on disease activity (clinical scales), quality of life, and lifestyle together with registry data on comorbidity and medication. During follow-up evaluation of a successful treatment outcome response will be based on clinical scales and most frequently used primary endpoints; the major outcome of the analyses will be to detect differences in treatment outcome between patients in different treatment group.

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of uni or bilateral uveitis
* recurrence of the diagnosed previously uni or bilateral uveitis

Exclusion Criteria:

* not mentally able to reply the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a new diagnosis or a recurrence of uni or bilateral uveitis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success | 1 year
  Total number of treatment success in each group
Recurrence time | 10 years
  Time to the next recurrence after the treatment regimen introduction
Severe visual loss | 10 years
  Time and cause of severe visual loss

SECONDARY OUTCOMES:
ETDRS Visual Acuity | 10 years
  Visual Acuity will be performed with ETDRS charts different for right and left eye
The SUN working group grading system for anterior chamber cells | 10 years
  At each visit anterior chamber will be examined to assess anterior chamber cells (1mm x 1mm slit beam in height and width, when thrown at an angle of 45-60°). The recorded number of cells will be used to determine the grade according to the SUN criteria.
The SUN working group grading system for anterior chamber flare | 10 years
  At each visit anterior chamber will be examined to assess anterior chamber flare (1mm x 1mm slit beam in height and width, when thrown at an angle of 45-60°). The observed changes will be used to determine the grade according to the SUN criteria.
AREDS 2008 Clinical Lens Opacity Grading Procedure | 10 years
  Using AREDS system for classifying cataracts from photographs: AREDS Report No. 4 the lens opacity will be graded.
NIH grading system for vitreous cells | 10 years
  At each visit vitreous will be examined to assess vitreous cells (1mm x 3mm slit beam in anterior vitreous). The recorded number of cells will be used to determine the grade according to the NIH criteria.
NIH grading system for vitreous haze | 10 years
  At each visit vitreous will be examined to assess vitreous haze. The recorded of clarity of posterior pole funduscopy will be used to determine the grade according to the NIH criteria.
Submacular choroidal thickness | 10 years
  OCT EDI recordings processed with developed by researchers methodology for image processing.

OTHER OUTCOMES:
COVID-19 confirmed infection asymptomatic patient | 1 year
  PCR-positive result of COVID-19 specific testing, no treatment required
COVID-19 confirmed infection | 1 year
  PCR-positive result of COVID-19 specific testing, patient require treatment. The mode of treatment will be recorded into several groups: 1) antibiotics, 2) antivirals, 3) biologic treatment, 4) immunoglobulins, 5) steroids
COVID-19 related acute respiratory distress syndrome (ARDS) | 1 year
  COVID-19 related acute respiratory distress syndrome (ARDS). Situation in which patients need any of described below: 1) supportive oxygen therapy, 2) non-invasive ventilation, 3) invasive/ mechanical ventilation, 4) use of ECMO, 5) admission to intensive care unit, 6) dialysis
Ocular Surface Disease Index | 1 year
  Ocular Surface Disease Index (OSDI) questionaire results are used to define if during the course of the disease the dry eye syndrom occurs. Used with subclasses describing the vision-related functions, ocular symptoms, environmental triggers
Dry Eye Questionnaire | 1 year
  Dry Eye Questionnaire (DEQ 5) questionaire results are used to define if during the course of the disease the dry eye syndrom occurs. Used with subscales describing the eye dyscomfort, eye dryness and watery eyes.
SANDE Questionnaire | 1 year
  SANDE Questionnaire that assess the frequency and severity of symptoms during the treatment.
LIKERT Questionnaire | 1 year
  LIKER Questionnaire that assess the frequency, severity of symptoms and infuence of symptoms on the patient day-to-day activities during the treatment.
LIPCOF scale | 1 year
  Assesment of conjunctival folds according to pre-defined scale.
OXFORD scale | 1 year
  OXFORD scale conducted with instalation of 2 microliters of 2% fluorescite into the conjunctival sac and assessment according to the pre-defined scale. The subscales for nasal, temporal and lower lid conjunctiva as well as for cornea was used. The scale has been conducted during the treatment period and if necessary during additional visits.
SICCA scale | 1 year
  SICCA scale conducted with instalation of 2 microliters of 2% fluorescite into the conjunctival sac and assessment of cornea according to the pre-defined scale. Different dye was used for conjunctica (lizamine green). The subscales for nasal and temporal conjunctiva as well as for cornea was used. The scale has been conducted during the treatment period and if necessary during additional visits.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Misiuk-Hojło, Professor, Study Chair — Medical University of Wrocław
Locations (1):
- Department of Ophthalmology, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Sharing coded data such as BCVA, intraocular preassure, visual functioning questionaire responses, anterior chamber cells and flare scales records as well as lens opacity grading records.